CLINICAL TRIAL: NCT00004177
Title: Phase I/II Radioimmunotherapy With High-Dose 90Y-Labeled Humanized MN-14 in Advanced Ovarian Cancer Using Autologous Peripheral Blood Stem Cell Rescue (PBSCR) to Control Myelotoxicity
Brief Title: Radiolabeled Monoclonal Antibody Plus Peripheral Stem Cell Transplantation in Treating Patients With Refractory or Recurrent Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Garden State Cancer Center at the Center for Molecular Medicine and Immunology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert M Sharkey, GSCC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067299; R03CA077146 (NIH); CMMI-C-039A-98; NCI-H99-0044; NCI-V99-1570
Record Dates: First submitted 2000-01-21; First posted 2004-04-16 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Filgrastim; Peripheral Blood Stem Cell Transplantation; Indium

INTERVENTIONS:
Biological: filgrastim — as prescribed by physician
Procedure: peripheral blood stem cell transplantation — 1-2 weeks from treatment
Radiation: indium In 111 monoclonal antibody MN-14 — intravenous infusion over 30 min; single dose
Radiation: yttrium Y 90 monoclonal antibody MN-14 — intravenous infusion over 30 min; single dose

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by therapy used to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiolabeled monoclonal antibody plus peripheral stem cell transplantation in treating patients who have refractory or recurrent ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the normal organ and tumor dosimetry with yttrium Y 90 monoclonal antibody MN-14 using indium In 111 monoclonal antibody MN-14 as pretherapy in patients with advanced ovarian epithelial cancer. II. Evaluate the extent and duration of antitumor response in these patients on this regimen.

OUTLINE: This is a dose escalation study of yttrium Y 90 monoclonal antibody MN-14 (90Y hMN-14). Patients receive filgrastim (G-CSF) subcutaneously (SQ) on days -17 to -13, followed by leukapheresis on days -14 to -12. If an adequate number of CD34+ cells are not harvested, bone marrow is also collected. Patients receive pretherapy targeting consisting of indium In 111 monoclonal antibody MN-14 over 30 minutes on day -7. At least 1 confirmed tumor site must be targeted. Patients receive 90Y hMN-14 IV over 30-45 minutes on day 0. PBSC is reinfused within 7 to 14 days after 90 hMN-14 administration. Patients receive G-CSF SQ or IV until blood counts recover. Cohorts of 3-6 patients receive escalating doses of 90Y hMN-14 until the maximum tolerated dose (MTD) is determined. The MTD is defined as either the dose at which no more than 1 of 6 patients experiences dose limiting toxicity or the threshold radiation doses to lungs, kidney, and liver are reached. Patients are followed weekly for 1 month, every 2 weeks for 2 months, monthly for 3 months, every 3 months for 2 years, and then every 6 months for 5 years.

PROJECTED ACCRUAL: Approximately 48-51 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically refractory or recurrent ovarian epithelial cancer Resistant to platinum or taxane containing chemotherapy within past 6 months Autologous peripheral blood stem cells (PBSC) or bone marrow available At least 1 measurable site confirmed by CT targeted pretherapy indium In 111 monoclonal antibody MN-14 imaging No bone marrow involvement

PATIENT CHARACTERISTICS: Age: 18 to 80 Performance status: Karnofsky 70-100% ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT less than 2.0 times upper limit of normal (ULN) Renal: Creatinine less than 1.5 times ULN Creatinine clearance at least 50 mL/min Cardiovascular: LVEF at least 50% by MUGA Pulmonary: FVC, FEV1, and DLCO at least 70% of predicted Other: Not pregnant Fertile patients must use effective contraception during and for 3 months after study No AIDS-related illness No concurrent significant medical complications that would preclude compliance No severe anorexia, nausea, or vomiting No history of allergy or antibodies to 90Y hMN-14

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior imaging studies with murine monoclonal antibodies showing reactivity with yttrium Y 90 monoclonal antibody MN-14 (90Y hMN-14) Chemotherapy: At least 4 weeks since prior chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy to index lesion and recovered No prior radiotherapy to greater than 25% of red marrow No prior radiotherapy to maximum tolerated levels for any critical organ (e.g., lung, liver, or kidney) Surgery: At least 4 weeks since prior major surgery Other: No concurrent antiretroviral medication

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 1999-08; Primary Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jack D. Burton, MD, Study Chair — Garden State Cancer Center at the Center for Molecular Medicine and Immunology
Locations (3):
- United States (3):
  - Garden State Cancer Center, Belleville, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania